CLINICAL TRIAL: NCT07277283
Title: Time to Target Blood Pressure Before Reperfusion Therapy in Acute Ischemic Stroke: Nicardipine Versus Labetalol
Brief Title: Nicardipine vs. Labetalol
Acronym: AISstdy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 01-2025
Record Dates: First submitted 2025-11-22; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke; Hypertensive Crisis
Keywords: Acute ischemic stroke; Nicardipine; Labetalol; time to achievement of target blood pressure; door-to-needle time; early neurological improvement
MeSH Terms: conditions — Ischemic Stroke; Hypertensive Crisis

STUDY DESIGN:
Intervention Model Description: Single center
Who Masked: Investigator
Masking Description: Patients were randomly assigned to the nicardipine or labetalol groups using a web-based computer-generated randomization service (https://www.randomizer.org/). Allocation concealment was ensured using sequentially numbered, opaque, sealed envelopes (SNOSE). Envelopes were prepared and sealed according to the randomization list and opened sequentially after eligibility had been confirmed and written informed consent obtained.
  Clinicians administering the interventions were not blinded to treatment allocation but were not involved in outcome assessment or data analysis. Outcome assessors and the statistical team were blinded to treatment assignment. Treatment codes were accessible only in emergency safety situations requiring unblinding, and such cases were documented according to the study protocol. All primary analyses were conducted according to the intention-to-treat (ITT) principle, with per-protocol analyses reported as sensitivity analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nicardipine group (Active Comparator): The nicardipine group received an IV infusion of nicardipine.
  Interventions: Drug: nicardipine intravenous
- Labetalol group (Active Comparator): The labetalol group received an IV bolus of labetalol.
  Interventions: Drug: labetalol intravenous

INTERVENTIONS:
Drug: nicardipine intravenous — In the nicardipine group, an 18-gauge peripheral IV catheter was preferably placed in the antecubital fossa. Continuous infusion was initiated at a starting dose of 5 mg/hour and titrated upward by 1 mg/hour every 5 minutes according to the BP response. Administration was performed using an electronic infusion pump.
  Arms: Nicardipine group
Drug: labetalol intravenous — In the labetalol group, an 18-gauge peripheral IV catheter was preferably placed in the antecubital fossa. An initial 20 mg dose of labetalol was administered as an IV bolus. If needed, additional 20 mg boluses were given every 5 minutes, not exceeding a cumulative dose of 300 mg.
  Arms: Labetalol group

SUMMARY:
In this ED-based study, the investigators compared the time to reach target blood pressure (BP) between hypertensive patients with acute ischemic stroke (AIS) undergoing intravenous (IV) thrombolysis and/or mechanical thrombectomy who received IV nicardipine versus labetalol. Additionally, the investigators evaluated the rate of early neurological improvement (ENI), length of hospital stay (LOS), in-hospital mortality, and adverse event profiles between the two treatment groups.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a leading cause of death and long-term disability worldwide. In patients who are candidates for intravenous thrombolysis and/or mechanical thrombectomy, rapid and controlled reduction of markedly elevated blood pressure (BP) before reperfusion therapy is critical for both treatment success and safety. International guidelines recommend intravenous nicardipine and labetalol as first-line antihypertensive agents in this setting; however, existing evidence comparing these two strategies is heterogeneous, and there is ongoing uncertainty regarding which agent facilitates faster and more stable BP control in the pre-reperfusion phase.

This prospective, randomized, single-blind, single-center clinical trial evaluates two commonly used intravenous antihypertensive regimens-nicardipine versus labetalol-for BP management in hypertensive AIS patients presenting to the emergency department. Consecutive adult patients with a clinical and radiological diagnosis of AIS and severely elevated BP at presentation who were planned for reperfusion therapy were screened for eligibility.

After written informed consent was obtained, eligible patients were randomly allocated in a 1:1 ratio to receive either intravenous nicardipine or intravenous labetalol. Randomization was performed using a computer-generated sequence with allocation concealment (sequentially numbered, opaque, sealed envelopes). Treating clinicians were aware of group allocation in order to administer the assigned drug, whereas outcome assessors and the statistical team remained blinded throughout data collection and analysis.

In the nicardipine arm, patients received a continuous intravenous infusion via a peripheral venous catheter using an electronic infusion pump, with the dose titrated at short intervals according to BP response. In the labetalol arm, patients received intermittent intravenous bolus doses through a peripheral line, with repeated boluses permitted up to a predefined cumulative limit when needed. In both groups, continuous cardiac and hemodynamic monitoring was maintained during antihypertensive therapy. BP was measured at frequent, standardized intervals using automated devices and verified manually when indicated. Once the predefined BP target recommended for pre-reperfusion management in AIS was achieved, the study drug was down-titrated or withheld, and patients proceeded to reperfusion therapy in accordance with current stroke guidelines and local protocols.

Time from initiation of antihypertensive treatment to achievement of target BP is the main efficacy endpoint of this trial. Secondary endpoints include additional time-based metrics related to reperfusion therapy, drug exposure parameters, the occurrence of predefined cardiovascular and hemodynamic adverse events during antihypertensive treatment, early neurological response, and in-hospital clinical course. Neurological status is assessed using the National Institutes of Health Stroke Scale (NIHSS) at baseline and during early follow-up, and standard radiological imaging is used to identify treatment-related intracranial complications. All clinically relevant data are collected prospectively using a standardized case report form and analyzed according to an intention-to-treat approach.

This study is designed to generate prospective randomized data on the comparative effectiveness and safety of nicardipine and labetalol for pre-reperfusion BP management in hyperacute AIS. By focusing on time-to-target BP and short-term clinical outcomes in a real-world emergency department setting, the trial aims to inform clinicians' choice between these two widely used antihypertensive strategies in time-critical stroke care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presentation to the emergency department with clinical and radiological evidence of acute ischemic stroke (cranial CT with or without CT angiography, or diffusion-weighted MRI)
* Initial systolic blood pressure (SBP) ≥ 185 mmHg and/or diastolic blood pressure (DBP) ≥ 110 mmHg

Exclusion Criteria:

* Age < 18 years
* Intracranial hemorrhage, subarachnoid hemorrhage, or other non-stroke structural pathology on initial neuroimaging
* Stroke mimics (e.g., hypoglycemia, postictal paresis)
* Absolute contraindication to reperfusion therapy at presentation such that pre-procedural blood pressure control is not planned as part of clinical management
* Achievement of target blood pressure with prior antihypertensive treatment or receipt of other intravenous antihypertensive agents before randomization
* Hemodynamic instability or respiratory failure requiring emergency intubation and advanced life support
* Contraindications to labetalol or nicardipine (e.g., severe bronchospastic disease, advanced atrioventricular block, or critical aortic stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Time to reach target blood pressure | at 15 minutes after the drug administration
  The investigators assessed the time from the initiation of antihypertensive drug to the first confirmation of target BP (SBP ≤185 mmHg and DBP ≤110 mmHg).

SECONDARY OUTCOMES:
The proportion of patients achieving target BP | at 15 minutes after the drug administration.
  The investigators assessed the proportion of patients achieving target BP within the first 15 minutes.
Door-to-needle time | From emergency department admission to initiation of intravenous thrombolytic therapy, assessed up to 24 hours after emergency department arrival.
  The investigators assessed the door-to-needle time in patients with acute ischemic stroke.
The frequency and types of adverse events | from emergency room admission to the 24 hours.
  The investigators assessed the frequency and types of adverse events in acute ischemic stroke patients undergoing IV thrombolysis and/or mechanical thrombectomy who received IV nicardipine versus labetalol

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, Assoc. Prof., Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Result] Guo QH, Liu CH, Wang JG. Blood Pressure Goals in Acute Stroke. Am J Hypertens. 2022 Jun 16;35(6):483-499. doi: 10.1093/ajh/hpac039. PMID 35323883
- [Result] Huang A, Parker D Jr, Wein R. Comparison of nicardipine versus labetalol for time to alteplase administration in acute ischemic stroke. Front Neurol. 2025 Jul 2;16:1573352. doi: 10.3389/fneur.2025.1573352. eCollection 2025. PMID 40672455
- [Result] Hao F, Yin S, Tang L, Zhang X, Zhang S. Nicardipine versus Labetalol for Hypertension during Acute Stroke: A Systematic Review and Meta-Analysis. Neurol India. 2022 Sep-Oct;70(5):1793-1799. doi: 10.4103/0028-3886.359214. PMID 36352567
- [Result] Ortega-Gutierrez S, Thomas J, Reccius A, Agarwal S, Lantigua H, Li M, Carpenter AM, Mayer SA, Schmidt JM, Lee K, Claassen J, Badjatia N, Lesch C. Effectiveness and safety of nicardipine and labetalol infusion for blood pressure management in patients with intracerebral and subarachnoid hemorrhage. Neurocrit Care. 2013 Feb;18(1):13-9. doi: 10.1007/s12028-012-9782-1. PMID 23055089